CLINICAL TRIAL: NCT06651073
Title: Real-World Characteristics and Treatment Patterns of Patients With Transthyretin Amyloid Cardiomyopathy (ATTR-CM): A Multi-Country, Non-Interventional, Disease Registry
Brief Title: ATTR-CM: A Multi-country, Non-interventional Disease Registry
Status: Recruiting | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B3461110; NCT06651073 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2024-10-04; First posted 2024-10-21 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Transthyretin Amyloid Cardiopathy
Keywords: Transthyretin amyloid cardiopathy
MeSH Terms: interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ATTR-CM patients in Taiwan, Hong Kong, and Malaysia: case-only
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — There is no intervention involved in the study. It is purely observational.
  Other Names: Non-interventional, Observational

SUMMARY:
This study is a multi-center, non-interventional, disease registry to characterize the natural history of ATTR-CM and treatment patterns in clinically diagnosed ATTR-CM patients. Data will be collected in the course of routine clinical practice or following local standard practice guidelines. No procedures or treatments will be mandated by this study, patients will receive usual clinical care.

The patient population will include all adult patients with a confirmed diagnosis of ATTR-CM after 01 June 2019 and who meet eligibility criteria. The index date of each patient will be the date of the first documented ATTR-CM diagnosis. The observation period for each patient will range from the index date to whichever occurs first of death, patient withdrawal of consent, loss to follow-up, or end of data collection. The end of data collection (ie, the end of study) is planned for 12 months after the end of the enrollment period.

As this study is descriptive in nature with no hypothesis testing, the study size will be based on the number of eligible ATTR-CM cases identified in the medical records and meeting the eligibility criteria. Approximately 350 patients diagnosed with ATTR-CM across approximately 17 sites in Taiwan, Hong Kong, and Malaysia are planned to be enrolled.

DETAILED DESCRIPTION:
Study variables will include demographic and clinical characteristics of the ATTR-CM patients at diagnosis, including age, sex, physical measurement, relevant medical history and comorbidities, New York Heart Association (NYHA) functional class, prior prescription of heart and CV medication, type of ATTR-CM (ATTRwt or ATTRm), and diagnosis parameters. Exposure variables will include treatment type, treatment regimen/patterns, and concomitant medications. Outcome variables will provide information on death (status and reasons), hospitalizations (status and reasons), imaging and lab assessments, Kansas City Cardiomyopathy Questionnaire (KCCQ), and healthcare resource utilization (eg, days of hospitalization, frequency of emergency department visits). All relevant data will be collected from the index date to the end of the observation period.

Data will be obtained from all information that is available at the site in the patients' electronic medical records and medical charts (eg, consultation notes, discharge summaries, laboratory test results, recorded prescription data, and any other documentation of communication with other health care providers). All data will be collected by trained site personnel and entered directly into web-based electronic case report forms (eCRFs).

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the patient (or a legally acceptable representative) has been informed of all pertinent aspects of the study. Waivers of informed consent for deceased patients will be pursued if permitted by local regulation
2. Patients aged ≥18 years at first ATTR-CM diagnosis
3. Patients with confirmed diagnosis of ATTR-CM after 01 June 2019

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population will include all adult patients with a confirmed diagnosis of ATTR-CM after 01 June 2019 and who meet eligibility criteria. The index date of each patient will be the date of the first documented ATTR-CM diagnosis. The observation period for each patient will range from the index date to whichever occurs first of death, patient withdrawal of consent, loss to follow-up, or end of data collection. The end of data collection (ie, the end of study) is planned for 12 months after the end of the enrollment period.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-10-03 (Estimated); Study Completion 2025-10-03 (Estimated)

PRIMARY OUTCOMES:
Demographic data | From Enrollment/Baseline to 12 months
  Age (measured in years) at enrollment, sex/gender (male/female), race/ethnicity
Physical measurements (in all patients whether receiving treatment or not) | index date (closest available measurement) to 12 months
  Height (in cm), weight (in kg), smoking status (never/prior/current), blood pressure (diastolic/systolic [in mmHg], heart rate (in beats/minute)
Relevant medical history and comorbidities | enrollment/baseline to 12 months
  The following information will be collected: First clinical cardiac symptom related to ATTR-CM, symptom onset date, age at onset of symptom; treatment received for the first symptom (with start and end date); Relevant medical history and comorbidities of interest including: amyloidosis, CV conditions (HFpEF, HFrEF, left ventricular hypertrophy/increased wall thickness, ischemic heart disease, pulmonary embolism, pericarditis, aortic stenosis, cardiac arrhythmias, atrial fibrillation and flutter, atrioventricular and left bundle branch block, conduction disorders, pacemaker or implantable cardioverter-defibrillator, other) Other vascular comorbidities: hypertensive diseases, diabetes mellitus, cerebrovascular disease, peripheral vascular disease, venous thrombosis, other. Nervous system conditions: carpal tunnel syndrome, lumbar spinal stenosis, peripheral neuropathy, autonomic neuropathy, other. Genitourinary system conditions: chronic kidney disease, erectile dysfunction, other.
NYHA Functional Class | index date (closest available measurement to enrollment)
  Patients' Physical activities wil be graded I, II, III, IV. I being asymptomatic, II being slight limitation, III being marked limitation, and IV being symptoms at rest.
Prescription of heart and cardiovascular medication | within 6 months prior to the index date to 12 months
  The following information will be collected: Medication type (eg. beta-blockers, ACE inhibitors, ARBs, ARNi, digoxin, calcium channel blockers, diuretics, antiplatelets, lipid-lowering agents, anticoagulants, other), medication name, start date, end date, reason of discontinuation
Type of ATTR-CM | enrollment/index date
  described by whether it is wild type or hereditary (including genetic variant if identified)
Family History | index date/baseline
  Describe whether the patient has family history of known cardiomyopathy, polyneuropathy, and sudden cardiac death (among parents, siblings, and 2nd/3rd grade family)
Diagnosis of ATTR-CM | enrollment/baseline
  Date of first ATTR-CM diagnosis; Age (in years) at first ATTR-CM diagnosis; Method of diagnosis of ATTR-CM including any of the following: cardiological assessments, MRI, ECG, ECHO, PYP scan with SPECT/CT (for definite confirmatory testing), nerve conduction studies, plasma neurofilament light (pNfL), and any other methods

SECONDARY OUTCOMES:
Treatment for ATTR-CM | enrollment, every 3 month or as per standard of care, 12 months
  Type of Treatment including:
  1. ATTR-specific pharmacologic treatment: treatment name, dosage, frequency, start and end date, any treatment change, date and reason of treatment change.
  2. Supportive treatment of cardiac involvement: 1. management of HF; 2. management of arrhythmias: medical therapy (eg. rate/rhythm control, cardioversion/ablation, other), device therapy, and other.
  3. Liver or heart transplant.
  4. Other
Concomitant medications (including heart and CV medications and other concomitant medications) | from index date until 12 months
  The following information will be collected: Medication type (CV-related [eg. beta-blockers, ACE inhibitors, ARBs, ARNi, digoxin, calcium channel blockers, diuretics, antiplatelets, lipid-lowering agents, anticoagulants, or other] non-CV related), medication name, prescribed dose, dosing frequency, indication, start and stop dates, and reasons for discontinuation.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Lin YH, Chou HW, Tsai S, Gomez R. Real-World Characteristics and Treatment Patterns of Patients With Transthyretin Amyloid Cardiomyopathy: Protocol for a Multicountry Disease Registry Study. JMIR Res Protoc. 2025 Jun 6;14:e71314. doi: 10.2196/71314. PMID 40479720
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B3461110